CLINICAL TRIAL: NCT06474312
Title: A Randomized Controlled Trial to Examine the Feasibility, Relevance, and Effectiveness of the Tool "Nae Disha for Life" Module in Reducing Suicide Ideation Among Young People in Bundelkhand Region of Madhya Pradesh, India
Brief Title: Reducing Suicide Ideation Among Young People
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Christian Hospital Chhatarpur (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY23040073; 5D43TW009114-10 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Suicidal Ideation; Suicide, Attempted
Keywords: Nai Dish; Suicide ideation; Cue based; suicide attempts
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: The study is a Cluster Randomized Control Trial (CRCT) research / study. The selection and approval of 64 Government schools was obtained will be done by the local PI based on comparable demographics (i.e. similar levels of socio-economic status) in the Nowgong block of Chhatarpur district. Two of the four schools will receive the intervention (intervention arm) and the other two will be the control arm.
  A sample size of n = 170 young people in each arm will be recruited from participating schools who are studying in 7th and 8th classes, aged between 12 - 17 years old. Sample size was calculated using optimal design software.
  The demographic data (e.g. age, father and mother completed years of education, caste, religion, etc.) as well as psychometric measures will be collected at baseline (prior to intervention) and endline (post intervention).
  All participants below 18 years of age will only be recruited after parental consent and self-assent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Nae Disha (Experimental): "Nae Disha for Life" is a brief, multi-component, psychosocial promotion and resilience tool developed by Emmanuel Hospital Association, New Delhi. The purpose of this research work is to evaluate the feasibility, acceptance, and effectiveness of "Nae Disha for Life" tool in reducing suicide ideation among youth in Bundelkhand region. This will be implemented among the targeted schools of Nowgong block, Chhatarpur district.
  Interventions: Behavioral: Nae Disha
- Control arm (No Intervention): The control arm will not get any intervention,

INTERVENTIONS:
Behavioral: Nae Disha — "Nae Disha for Life" is a brief, multi-component, psychosocial promotion and resilience tool developed by Emmanuel Hospital Association, New Delhi. The purpose of this research work is to evaluate the feasibility, acceptance, and effectiveness of "Nae Disha for Life" tool in reducing suicide ideation among youth in Bundelkhand region. This will be implemented among the targeted schools of Nowgong block, Chhatarpur district.
  Arms: Intervention Nae Disha

SUMMARY:
It is Cluster Randomized Control Trial research to examine feasibility and relevance of the modified tool Nae Disha for Life, which will incorporate suicide prevention and resilience to reduce suicide ideation among young people in Bundelkhand region of Madhya Pradesh, India. This intervention will build on existing relationships with at least four Government Middle Schools in Nowgong block of Chhatarpur district, Madhya Pradesh. This preliminary research will develop relationships and evidence for implementation scale-up research.

DETAILED DESCRIPTION:
Madhya Pradesh state in India was ranked as third highest number of suicides reported in 2020 in India. The majority of suicide victims (23.4%) (35,771) were educated up to Matriculation/ Secondary level. A large proportion of suicide deaths occur between the ages 15 and 29. Mental health problems begin during youth (12-24) years of age, however, is often detected later in life.

"Nae Disha for Life" is a brief, multi-component, psychosocial promotion and resilience tool developed by Emmanuel Hospital Association, New Delhi. The purpose of this research work is to evaluate the feasibility, acceptance, and effectiveness of "Nae Disha for Life" tool in reducing suicide ideation among youth in Bundelkhand region. This will be implemented among the targeted schools of Nowgong block, Chhatarpur district.

There are number of studies on treatment gaps for the mental health problems, suicide statistical analysis, methods of suicides, and causes of suicides. But there is hardly any study on prevention of suicides or suicidal ideation among the youth in India.

However, Nae Disha is a youth resilience group-based intervention building on the Ottawa health promotion charter, that aims to increase and strengthen key psycho-social assets in adolescents to moderate the impacts of adversity. It has been successfully implemented amongst out-of-school adolescents in Northern India and studies have demonstrated effectiveness in improving perceptions of social inclusion, attitudes to gender equality, resilience, and mental health among young people affected by mental illness. The Nae Disha would also deliver benefits to other young people similarly affected in other parts of India, and possibly beyond.

Building on these studies, I propose to examine feasibility and relevance of the modified tool Nae Disha for Life, which will incorporate suicide prevention and resilience to reduce suicide ideation among young people in Bundelkhand region of Madhya Pradesh. This intervention will build on existing relationships with at least four Government Middle Schools in Nowgong block of Chhatarpur district, Madhya Pradesh. This preliminary research will develop relationships and evidence for implementational scale-up research.

The research activities of the study is distributed as follows:

4 months(16weeks), Training of surveyors, Training staff as Facilitators, Meeting with local, stakeholders / communities, Refinement of program content.

Next two weeks:Recruiting of subjects from 4 schools, Screening of subjects in 4 schools, Formation of groups in 4 schools,Baseline data collection from subjects,

18 weeks (Week 17-to week 34):Intensive implementation in intervention arm and control arm in 4 schools 2 (Week 35-36) weeks:Endline quantitative and qualitative data collection 6 weeks(week 37-week:43) Data entry, analysis and presentation of data findings After week 43: Dissemination meetings to be held at in schools and Chhatarpur

ELIGIBILITY:
Inclusion Criteria:

* Students of 7th and 8th classes of selected schools between 12 - 17 years old age group,

Exclusion Criteria:

* a. Students who are planning to move to other schools during intervention period

  b. Students of 7th/8th grade who turn 18 during the study.

  c. Those with chronic debilitating diseases or disorders who cannot participate in Nae Disha activities such as heart disease, epilepsy, cystic fibrosis, cerebral palsy, and any other diseases that the doctor has restricted the student to participate in it.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 272 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Suicide ideation | Baseline and after 18 weeks of intervention
  To study change in suicide ideation in intervention group measured by Beck Suicidal Ideation Scale as compared to control group. The total score ranges from 0 to 38.More score means higher suicide ideation.
Hopelessness | Baseline and after 18 weeks of intervention
  To study change in hopelessness in intervention group measured by Beck Hopelessness Scale as compared to control group. The score ranges from 0 to 20.
Generalized anxiety | Baseline and after 18 weeks of intervention
  To study change in generalized anxiety in intervention group measured by Generalized Anxiety Disorder Scale as compared to control group
Resilience | Baseline and after 18 weeks of intervention
  To study change in resilience in intervention group measured by Connor-Davidson Resilience Scale as compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, Principal Investigator — University of Pittburgh
Locations (1):
- Christian Hospital, Mahoba Road, Chhatarpur, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study
Access Criteria: For individual participant data, meta-analysis